CLINICAL TRIAL: NCT03225664
Title: A Biomarker-Integrated Targeted Therapy Study in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer - (IM-BATTLE-2 Program)
Brief Title: Trametinib and Pembrolizumab in Treating Patients With Recurrent Non-small Cell Lung Cancer That Is Metastatic, Unresectable, or Locally Advanced
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0226; NCI-2018-01107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0226 (Other: M D Anderson Cancer Center); R01CA155196 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Pharmacogenomic Variants; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trametinib, pembrolizumab) (Experimental): Patients receive trametinib PO QD 14 days prior to cycle 1 and days 1-10 of each course (10 days on, 11 days off). Beginning in cycle 2, participants also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Other: Pharmacokinetic Study; Drug: Trametinib

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of trametinib when given together with pembrolizumab and to see how well they work in treating patients with non-small cell lung cancer that has come back and spread to other places in the body, cannot be removed by surgery, or spread to nearby tissues or lymph nodes. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving trametinib and pembrolizumab may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity profile of trametinib, a MEK inhibitor, in combination with pembrolizumab, an anti PD-1 monoclonal antibody, as treatment for refractory to chemotherapy KRAS mutation positive (mut+) and KRAS wild-type patients with advanced non-small cell lung cancer (NSCLC) and establish a recommended dose for the combination for the phase II portion of the study. (Part 1) II. To determine the 6-month overall response rate (ORR) for the combination of trametinib + pembrolizumab in subjects with NSCLC who received prior cytotoxic chemotherapy and anti-PD1 or anti-PD-L1 therapy. (Part 2)

SECONDARY OBJECTIVES:

I. To evaluate overall response rates (ORRs) using modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1 and immune related [ir]RECIST) and duration of response (DOR), median progression free survival (PFS) and overall survival (OS) in KRAS mut+, KRAS wild-type, PD-L1+ and PD-L1 negative cohorts of patients.

II. To evaluate ORRs by immune-related RECIST (irRECIST). III. To assess the safety and tolerability of pembrolizumab in combination with trametinib at the recommended dose to be used in future studies.

IV. To characterize the pharmacokinetics of trametinib and pembrolizumab when administered in combination.

V. To identify prognostic and predictive markers for the two treatment regimens by analyzing pre- and on-treatment tumor biopsies.

EXPLORATORY OBJECTIVES:

I. Evaluate exploratory genomic and gene expression biomarkers and their relationships in tumors in response to study treatment.

II. Analyze circulating soluble factors including cytokines, chemokines, and antibodies against tumor and self antigens in response to clinical outcomes.

III. Assess the activation state, quantity, and phenotype of T cells, B cells, and natural killer cells and the presence of immune regulatory cells (myeloid-derived suppressor cells) (MDSC) in response to treatment.

IV. Examine changes in the localization and numbers of tumor infiltrating lymphocytes (TILs) expressing key markers (PD-1, CD8, CD4, CD45RO, granzyme, CD68, Foxp3) by immunohistochemistry in response to treatment.

V. Perform immune monitoring studies in tissue and blood and correlate with genomic profiling and outcomes including toxicities.

VI. Evaluate KRAS-mutation specific T cell response in patients before and after monotherapy with PEMBROLIZUMAB and the combination of PEMBROLIZUMAB and trametinib.

VII. Evaluate immunophenotypes within the context of subsets of KRAS co-mutations (KRAS/p53, KRAS/LKB1, KRAS/CDKN2A/B inactivation).

VIII. Collect and store archival diagnostic tumor samples, matched pre- and post-treatment tumor biopsy samples and deoxyribonucleic acid (DNA) (from tumor and blood) for future exploratory research into genes/genetic variation and factors that may influence resistance and/or sensitivity, and/or response to trametinib and/or PEMBROLIZUMAB.

IX. Explore the relationship between pharmacokinetic (PK) plasma trametinib levels, trametinib exposure, safety and clinical outcome measures.

X. Isolate peripheral blood mononuclear cells (PBMCs) from whole blood to enable flow cytometric analysis of additional markers and perform functional testing for antigen specificity and responsiveness, and T cell receptor (TCR) diversity.

XI. Perform flow cytometric analyses in tumor tissue. XII. Analysis of the host microbiome from stool. XIII. Analysis of micro ribonucleic acid (miRNA) platelets and analysis in response to study treatment.

OUTLINE: This is a phase Ib, dose-escalation study of trametinib followed by a phase II study.

Patients receive trametinib orally (PO) once daily (QD) 14 days prior to cycle 1 and days 1-10 of each course (10 days on, 11 days off). Beginning in cycle 2, participants also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic or unresectable, locally advanced, recurrent NSCLC that has been previously treated (subjects who have failed adjuvant or locally advanced therapy within 6 months are also eligible to participate in the study)
* The subject has biopsy accessible tumor and is willing to undergo biopsy prior to planned protocol treatment
* Confirmation of the presence or absence of EGFR mutations and ALK gene fusions prior to study enrollment in all subjects except for patients with histologies other than adenocarcinoma and NSCLC, not otherwise specified (NOS), as the frequency of these alterations is exceedingly rare in this histology. Subjects with known EGFR sensitizing mutational status or ALK fusion must have been treated and progressed on EGFR TKIs or ALK-directed therapy, or with tumors harboring EGFR T790M mutation to have received and progressed on therapy directed at the T790M mutation (e.g. osimertinib). Subjects with known ROS1 translocation must have been treated and progressed on ROS1-directed therapy
* Measurable disease according to RECIST 1.1 and irRECIST. At least one lesion of at least 1.0 cm in the long-axis diameter for a non-lymph node or at least 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 and irRECIST using either computed tomography (CT) or magnetic resonance imaging (MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of at least 1.5 cm
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L or at least 1500/mm^3 or at least 1.5 x 10^9/L
* Platelet count at least 100,000/mm^3 or at least 100 x 10^9/L
* Hemoglobin (Hb) at least 9 g/dL (or 5.69 mmol/L) at baseline (blood transfusions, hematopoietic growth factors and hematinics are not allowed during the 7 days prior to screening to correct Hb values less than 9 g/dL)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or >= 60 mL/minute for subjects with creatinine levels > 1.5 x the institutional ULN
* Serum total bilirubin =< 1.5 x ULN or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN except for subjects with liver metastases (mets) for whom ALT and AST should be =< 5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated PTT (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulant
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female and male subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol
* Patients must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Prior MEK inhibitor therapy is allowed
* Prior anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) is required for phase 2 part of the study. Subjects must be resistant (at least stable disease at 12 weeks of treatment with anti-PD1, anti-PD-L1 therapy) (cohort A) or refractory (progression within 12 weeks of starting anti-PD1 therapy) (cohort B) to an Food and Drug Administration (FDA) approved anti PD 1/PD L1 monoclonal antibody (mAb) as either monotherapy or in combination with other approved checkpoint inhibitors or other therapies according to their label, defined as (subjects must meet all of the following criteria):

  * Have received at least 2 doses of anti PD 1/PD L1 mAb
  * Progressive disease after anti PD 1/PD L1 mAb defined according to RECIST 1.1
  * Have documented progressive disease (PD) within 12 weeks of the last dose of anti PD 1/PD L1 mAb. Patients who were re-treated with anti PD 1/PD L1 mAb and patients who were on maintenance with anti PD 1/PD L1 mAb will be allowed to enter the trial as long as there is documented PD within 12 weeks of the last treatment date (with anti PD 1/PD L1 mAb)

    * Note - Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of that treatment and precluding retreatment with the same agent before progression of disease will also be eligible

Exclusion Criteria:

* Subjects participating in or who have participated in a study of an investigational agent or is using an investigational device within 4 weeks of the first dose of study treatment or have received any anti-cancer therapy, platinum-based chemotherapy, targeted, biological (including humanized antibodies), investigational, immunotherapy, or hormonal agent, within 4 weeks of the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had prior monoclonal antibody therapy within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Has received previous treatment with an immunomodulatory therapy (eg, anti PD 1/PD L1 or CTLA-4 agent) and was discontinued from that therapy due to a grade 3 or higher immune-related adverse event (irAE)
* Had prior chemotherapy, targeted small molecule therapy within 4 weeks, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from AEs due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if a subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
  * Note: patients who have received > 30 Gy to the thorax must have completed this radiation 6 months prior to enrollment in the study
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell and squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis, or has history of pneumonitis that required systemic corticosteroids for recovery
* Has an active infection requiring systemic therapy
* Has symptomatic ascites or pleural effusion. A subject who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the study, or in the opinion of the investigator, is not in the best interest of the subject to participate
* Has known psychiatric or substance abuse disorders that could interfere with cooperation with the requirements of the protocol
* Is pregnant or breastfeeding, or expecting to become pregnant or father a child within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study drug
* Has a known history of human immunodeficiency virus (HIV) (HIV ½ antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative]) is detected
* Has received a live vaccine within 30 days prior to the first dose of study drug
* History or current evidence/risk of retinal vein occlusion (RVO)
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval if that treatment cannot be either discontinued or switched to a different medication (not known to affect QT interval) prior to cycle 1 day 1 (C1D1)
* Any of the following cardiac abnormalities or history: a) clinically significant abnormal 12-lead electrocardiogram (ECG), QT interval (QT corrected by Bazett's formula [QTCB]) > 480 ms, b) inability to measure QT interval on ECG, c) personal or family history of long QT syndrome, d) implantable pacemaker or implantable cardioverter defibrillator, e) resting bradycardia < 55 beats/min, f) history or evidence of current clinically significant uncontrolled arrhythmias. Exception: subjects with controlled atrial fibrillation for > 30 days prior to randomization are eligible, g) history of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting, within 6 months prior to randomization, h) history or evidence of current >= class II congestive heart failure as defined by New York Heart Association (NYHA), i) treatment refractory hypertension defined as a blood pressure of systolic > 140 mm Hg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy, j) cardiac metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall objective response rate evaluated according to modified Response Evaluation Criteria in Solid Tumors (RECIST 1.1 and immune related [ir]RECIST) | At 6 months
  Each patient will have the KRAS mutation and PD-L1 status determined prior to treatment in order for stratified randomization. A futility monitoring will be carried out continuously to each stratum within each treatment arm after the primary endpoints of 6 patients have been observed in the corresponding marker groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinandos Skoulidis, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org